CLINICAL TRIAL: NCT03354000
Title: Engaging Diverse Patients in Using an Online Patient Portal
Brief Title: An RCT of an Online Training for Vulnerable Patients to Use an Online Patient Portal Website
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Courtney Lyles, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5R00HS022408-05 (AHRQ)
Record Dates: First submitted 2017-11-09; First posted 2017-11-27 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Electronic Health Records; Chronic Disease; Health Literacy
Keywords: Patient Portal; Healthcare disparities; Safety net healthcare system
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take-home online training (Placebo Comparator): Participants received a link to access the online tutorial videos on their own.
  Interventions: Behavioral: Take-home online training
- In-person online training (Active Comparator): Participants received an in-person tutorial of how to use the patient portal website with a trained research assistant.
  Interventions: Behavioral: In-person online training

INTERVENTIONS:
Behavioral: Take-home online training — We randomized patients to receive a link to access the online tutorial on their own. Participants in the take-home arm were given a paper handout with a link to the training materials and an outline of the steps for accessing the training curriculum.
  Arms: Take-home online training
Behavioral: In-person online training — For participants randomized to the in-person training arm, a trained research assistant prompted participants to log into the learning platform and guided them in accessing the training materials for portal features that were of interest to them. The staff member provided further explanation or clarification if participants had questions about the training material.
  Arms: In-person online training

SUMMARY:
Online patient portals are becoming ubiquitous in the US. Previous research has documented substantial usability barriers, especially among patients with limited health literacy. This pilot randomized pilot trial had the goal of determining the effectiveness of an in-person training with a scalable online video-based training program to increase portal use among patients in a safety net healthcare setting.

DETAILED DESCRIPTION:
The intervention in this study was a patient portal training curriculum with simple instructions and 11 how-to videos for accessing features of an online patient portal. Using a deeply participatory approach, this curriculum was created in consultation with a patient advisory board from the San Francisco Health Network, a local Medicaid health plan. From June until October 2016, 93 patients with 1 or more chronic diseases were randomized to receive either: 1) an in-person tutorial with a trained research assistant versus 2) a link to view the videos on their own. The primary outcome was portal log-in (yes/no) between 3 and 6 months post-training, assessed through a portal administrative dashboard within the EHR. Secondary outcome included baseline and follow-up survey measures on participants' perceptions of the portal use and their care, as well as views of the web-based lessons.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking as portal is only available in English
* diagnosed with at least one chronic condition

Exclusion Criteria:

* cognitive impairment
* visual impairment
* severe mental health conditions
* any circumstances that would make participation in the study difficult
* no previous email use
* self-reported usage of MYSFHEALTH

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Portal log-ins | 3-6 months post-training
  Logging into the portal website in the 3-6 months post-training (yes/no)

SECONDARY OUTCOMES:
eHealth Literacy | 3-6 months post-training
  The eHEALS is a measure of eHealth literacy developed to measure consumers' combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems. eHEALS was measured at baseline and follow-up via surveys
Portal sign-up | 3-6 months post-training
  Initiating sign-up process for the portal website (yes/no), as pulled from EHR chart review
Digital literacy skills | 3-6 months post-training
  Confidence in having skills to be able to use online portal website (scored from 1 to 0), as self-reported via baseline and follow-up surveys

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Lyles, PhD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- See also: Published paper summarizing trial findings - A Randomized Trial to Train Vulnerable Primary Care Patients to Use a Patient Portal — http://www.jabfm.org/content/32/2/248